CLINICAL TRIAL: NCT04663230
Title: Right Atrial Fibrosis in Pulmonary Hypertension
Acronym: RAFE-PH
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Sponsor
Other Study IDs: AZ 12320
Record Dates: First submitted 2020-11-09; First posted 2020-12-10 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Hypertension; Chronic Thromboembolic Pulmonary Hypertension; Pulmonary Arterial Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pulmonary arterial hypertension: Patients with mean pulmonary arterial pressure above 25 mmHg, and a pulmonary capillary wedge pressure below 15 mmHg classified into group 1 of the clinical classification of pulmonary hypertension.
  Interventions: Diagnostic Test: cardiac magnetic resonance imaging
- Chronic thromboembolic pulmonary hypertension: Patients with mean pulmonary arterial pressure above 25 mmHg, and a pulmonary capillary wedge pressure below 15 mmHg with a history of pulmonary embolism, classified into group 4 of the clinical classification of pulmonary hypertension.
  Interventions: Diagnostic Test: cardiac magnetic resonance imaging
- Control: Patients with invasive exclusion of pulmonary hypertension (mean pulmonary arterial pressure below 25 mmHg) undergoing diagnostic CMRI due to the evaluation of dyspnoea.
  Interventions: Diagnostic Test: cardiac magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: cardiac magnetic resonance imaging — right atrial late gadolinium enhancement in % and cm2

SUMMARY:
The study aim to assess right atrial (RA) remodeling, in terms of RA fibrosis, in pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension patients. This will be investigated in detail with in-depth cardiac magnet resonance imaging (CMRI). A cohort with exclusion of pulmonary hypertension which underwent CMRI due to dyspnoe of unkown reason will be the control group.

DETAILED DESCRIPTION:
Right atrial (RA) function consists of a reservoir, conduit, and active contractile function and can serve as a tool for the evaluation of the severity of RV dysfunction and prognosis in pulmonary hypertension according to recent data. In-depth evaluation of phasic RA function was previously undertaken either by echocardiographic speckle tracking or by cardiac magnetic resonance (CMR) imaging-derived feature tracking. However, it is currently unknown if right atrial remodeling is present.

As described for left atrial fibrosis, the presence and extent of atrial fibrosis can be quantified using CMR late gadolinium enhancement. The protocol for the assessment of left atrial fibrosis will be used and adapted to the RA. Patients will undergo 3-dimensional late gadolinium enhancement CMRI along with a contrast-enhanced magnetic resonance angiography and cine imaging in order to define the anatomy of the RA and the superior and inferior vein. High-resolution late gadolinium enhancement images of the RA will be acquired 15 to 30 min after gadolinium-based contrast agents administration using a 3-dimensional inversion-recovery prepared, respiration navigated, and electrocardiogram triggered gradient-echo pulse sequence with fat saturation. Following acquisition of the scans, the endocardial borders of the RA will be defined in each slice by manual tracing. After manual adjustment of the epicardial RA surface, the quantification of fibrosis based on the relative intensity (signal intensity) of late gadolinium enhancement will be performed. Finally, a 3-dimensional model of the RA will be rendered with the maximum enhancement intensities being projected on the model surface.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of pulmonary arterial hypertension, WHO group 1 or chronic thromboembolic pulmonary hypertension, group 4
* Invasive exclusion of pulmonary hypertension
* Age ≥ 18 years
* Signed informed consent
* planned right heart catheterization based on clinical grounds

Exclusion Criteria:

* Other etiologic groups of pulmonary hypertension (WHO group 2, 3, 5)
* Patients with congenital heart disease
* Atrial septal defects
* Clinical relevant left heart disease
* Atrial fibrillation / Atrial flutter
* Ablations of the right atrium
* History of major cardiac surgery
* Atrial occlude
* Metallic implants
* Pacemakers
* Severe renal impairment (eGFR < 30 ml/min)
* Other severe disease with a life expectancy below 12 month
* Pregnancy
* Any known factor or disease that might interfere with treatment compliance, study conduct, or interpretation of results
* Intolerance to a contrast agent containing gadolinium
* Inability to perform a cardiac magnetic resonance imaging (claustrophobia or similar)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 subjects with pulmonary arterial hypertension, group 1 and chronic thromboembolic pulmonary hypertension, group 4; Patients with invasive exclusion of pulmonary hypertension undergoing diagnostic right heart catheterisation due to dyspnoe will serve as control
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
atrial fibrosis | 1 day
  right atrial late gadolinium enhancement in % and cm2

SECONDARY OUTCOMES:
Correlation of right atrial fibrosis with functional and exercise capacity | 1 day
  right atrial late gadolinium enhancement in % and cm2 correlated with 6minute walking distance in m or peak oxygen uptake in ml/min/kg
Correlation of right atrial fibrosis with remodeling of the right atrium, backflow and systemic congestion | 1 day
  right atrial late gadolinium enhancement in % and cm2 correlated with right atrial size (volume and cm2) and inferior vena cava diameter in cm2
Correlation of right atrial fibrosis with pulmonary hemodynamics | 1 day
  right atrial late gadolinium enhancement in % and cm2 correlated with mean right atrial pressure
Correlation of right atrial fibrosis with load-independent right ventricular function assessed by pressure-volume loop catheterization | 1 day
  right atrial late gadolinium enhancement in % and cm2 correlated with end-systolic to arterial elastance
Correlation of right atrial fibrosis with biomarkers | 1 day
  right atrial late gadolinium enhancement in % and cm2 correlated with B-type natriuretic peptide in pg/ml
Prognostic relevance of right atrial fibrosis | 1 day
  right atrial late gadolinium enhancement in % and cm2 as a predictor of clinical worsening or death

CONTACTS AND LOCATIONS:
Overall Officials: Richter Manuel, MD, Principal Investigator — UKGM Giessen
Locations (2):
- Germany (2):
  - Kerckhoff-Klinik, Bad Nauheim, Hesse
  - University of Giessen, Giessen, Hesse

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request